CLINICAL TRIAL: NCT01043471
Title: The Effects of Gum Chewing on Energy Intake and Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: The Obesity Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2007-0342
Record Dates: First submitted 2009-12-15; First posted 2010-01-06 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Chewing Gum; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chewing gum (Experimental)
  Interventions: Other: Chewing gum
- Water (Placebo Comparator)
  Interventions: Other: Water

INTERVENTIONS:
Other: Chewing gum — Subjects were instructed to chew gum at least 6 times a day in an effort to reduce snacking.
  Arms: Chewing gum
Other: Water — Subjects were instructed to drink 8 oz of water at least 6 times a day in an effort to reduce snacking.
  Arms: Water

SUMMARY:
The purpose of this study is to determine if chewing gum increases energy expenditure and decreases food intake.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-37, between the ages of 18 and 38

Exclusion Criteria:

* History of chronic disease (e.g. liver, kidney, or heart disease, or diabetes)
* Medications that affect energy expenditure, appetite, or body composition (e.g. antidepressants, beta blockers, antipsychotic, or weight loss medications)
* A history of irregular menstrual cycles in women (indication of onset of menopause or other metabolic disturbances such as polycystic ovary syndrome)
* A history of phenylketonuria (PKU)
* Symptoms of depression
* A history of eating disorders
* Concurrent participation in a weight loss program
* Cigarette smoking or other tobacco use
* Jaw problems such as temporomandibular joint disorder (TMJ)
* Allergies to any of the common components in gum (sweeteners, mint flavors, etc)
* Heavy gum chewing prior to study ( > 3 times per week)
* Pregnancy or lactation.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2008-09; Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Change in body composition | Baseline and end of study (6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Leah D Whigham, PhD, Principal Investigator — Board of Regents of the University of Wisconsin System
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States